CLINICAL TRIAL: NCT05526859
Title: Effect of Wrist Flexors Inhibition in Comparison to Wrist Extensors Facilitation Through Kinesiotaping Technique in Chronic Hemiplegic Stroke Patients With Limited Wrist Extension
Brief Title: Effect of Kinesiotape Technique on Wrist Among Chronic Stroke Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shifa Tameer-e-Millat University (Other)
Responsible Party: Principal Investigator, Nouman Khan, Lecturer, Shifa Tameer-e-Millat University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Saman IRB00
Record Dates: First submitted 2022-08-31; First posted 2022-09-02 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-08

CONDITIONS: Chronic Stroke
Keywords: Stroke; Manual Muscle testing; Kinesiotape; Range of Motion; Upper Extremity Functional Index; Modified Ashworth Scale
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Two group were taken and given treatment with the concern study protocols.
Who Masked: Participant
Masking Description: The participants were blinded to the allocation in the experimental treatment groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Hyperactive muscle correction for wrist extensors: Kinesiotape was applied to facilitate wrist extensor muscles from proximal to distal with 15-35% tension in therapeutic zone and no tension at anchor and end.
  Interventions: Other: Kinesiotaping for wrist extensor muscles
- Group 2 (Experimental): Hypoactive muscle correction for wrist flexors: Wrist flexors muscles were inhibited by applying tape from distal to proximal with 15-25% tension in therapeutic zone and no tension at anchor and end.
  Interventions: Other: Kinsiotaping for wrist flexor muscles

INTERVENTIONS:
Other: Kinsiotaping for wrist flexor muscles — The flexor muscles of the wrist area will be targeted.
  Arms: Group 2
Other: Kinesiotaping for wrist extensor muscles — The extensor muscles of the wrist area will be targeted.
  Arms: Group 1

SUMMARY:
The aim of this randomized controlled is to assess the effect of kinesiotape technique upon wrist joint among the patients with chronic stroke. Patients are devided into groups, in group A kinesiotaping facilitation technique is applied on wrist extensor muscles while inhibition technique is applied on wrist flexor muscles and the result is the compared between the groups and within the group.

DETAILED DESCRIPTION:
Stroke is a very common disease worldwide causing severe musculoskeletal disability due to which quality of life of patient compromises, patient becomes dependent of assistance in daily living activities and few becomes bed ridden. Stroke also causes death of the patient. Apart from musculoskeletal issues patient's cognitive abilities are also effected. It is tough to manage these patients as stroke varies in types and symptoms. Symptoms and severity depend upon type of stroke and factors like lifestyle, age and health issues. According to the symptoms different physiotherapy techniques and rehabilitation is used along with medical treatment and counseling of the patient. Kinesiotape also has the advantage that it can be worn 3-5 days due to which it's effects remains for long time as compare to other treatments which are given and has effect for a specific time for example a session of physical therapy including exercises is for an hour but this tape can be worn for days once applied.

Randomized controlled trial was done, 24 patients were recruited according to inclusion exclusion criteria. Patients were further divided into two groups; group 1 was given muscular facilitation treatment for wrist extensors and group 2 was given sessions for muscle inhibition treatment for wrist flexors. 6 sessions were given, 1 session per week over the period of 6 weeks to each patient.

Wrist range of motion for extension, flexion, ulnar and medial deviation was measured using goniometer before and after the 6 weeks. Manual muscle test for wrist extensors, modified ashworth scale and upper limb functional index scoring was done before and after sessions. Data was collected from a private clinic of PWD Rawalpindi.

The statistical values of result showed no significant change in between both the groups, before and after treatment. But a significant improvement was about observed within the group analysis It can be concluded from this study that Kinesiotape is an effective treatment method both in inhibiting and facilitating muscular performance. Hence both treatments were equally effective. it helps in increasing range of motion and in reducing spasticity.

ELIGIBILITY:
Inclusion Criteria:

* Age b/w 40 to 90
* Limited ROM (wrist extension)

Exclusion Criteria:

* Disoriented
* Who needs more then moderate support to achieve basic ADL and are bed bound
* Communication gap
* Allergic to Kinesiotaping after being positive to patch test

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-08-31 (Actual); Primary Completion 2022-10-19 (Estimated); Study Completion 2022-10-26 (Estimated)

PRIMARY OUTCOMES:
Wrist extensors manual muscle test score | 6 weeks
  Wrist extensors strength was measured as baseline before the start of intervention and was compared with the measurement after 6 weeks of application of kinesiotape.
Wrist ROMS through Goniometer | 6 weeks
  Wrist ROM was measured using universal goniometer, baseline values for wrist flexion, extension, ulnar deviation and medial deviation was measured and then compared to the values measured after 6 weeks of intervention.
Spasticity through modified ashwoth scale | 6 weeks
  Wrist spasticity was measured through modified ashworth scale before the intervention and then was compared with the values taken after 6th week
Upper extremity functional index (UEFI) | 6 weeks
  Patient was asked to perform different activities as opening the door and combing hair, score was done according to the difficulty level faced by patients while performing the activities. Measurement was taken before first session and was compared with the values taken after 6 weeks of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Saman Tauseef, MSPT, Principal Investigator — Shifa Tameer-e-Millat University
Locations (1):
- Shifa Tameer-e-Millat University, Islamabad, Fedral, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Akpalu J, Akpalu A, Ofei F. The metabolic syndrome among patients with cardiovascular disease in Accra, Ghana. Ghana Med J. 2011 Dec;45(4):161-6. PMID 22359422
- [Background] Anwar A, Saleem S, Aamir A, Diwan M. Organization of Stroke Care in Pakistan. Int J Stroke. 2020 Jul;15(5):565-566. doi: 10.1177/1747493019879663. Epub 2019 Sep 30. PMID 31564238
- [Background] Bernhardt J, Hayward KS, Kwakkel G, Ward NS, Wolf SL, Borschmann K, Krakauer JW, Boyd LA, Carmichael ST, Corbett D, Cramer SC. Agreed definitions and a shared vision for new standards in stroke recovery research: The Stroke Recovery and Rehabilitation Roundtable taskforce. Int J Stroke. 2017 Jul;12(5):444-450. doi: 10.1177/1747493017711816. PMID 28697708
- [Background] Cramer SC. Repairing the human brain after stroke: I. Mechanisms of spontaneous recovery. Ann Neurol. 2008 Mar;63(3):272-87. doi: 10.1002/ana.21393. PMID 18383072
- [Background] Drouin JL, McAlpine CT, Primak KA, Kissel J. The effects of kinesiotape on athletic-based performance outcomes in healthy, active individuals: a literature synthesis. J Can Chiropr Assoc. 2013 Dec;57(4):356-65. PMID 24302784
- [Background] Huang YC, Chang KH, Liou TH, Cheng CW, Lin LF, Huang SW. Effects of Kinesio taping for stroke patients with hemiplegic shoulder pain: A double-blind, randomized, placebo-controlled study. J Rehabil Med. 2017 Mar 6;49(3):208-215. doi: 10.2340/16501977-2197. PMID 28233009
- [Background] Kwakkel G, Kollen BJ, van der Grond J, Prevo AJ. Probability of regaining dexterity in the flaccid upper limb: impact of severity of paresis and time since onset in acute stroke. Stroke. 2003 Sep;34(9):2181-6. doi: 10.1161/01.STR.0000087172.16305.CD. Epub 2003 Aug 7. PMID 12907818
- [Background] Naci B, Ozyilmaz S, Aygutalp N, Demir R, Baltaci G, Yigit Z. Effects of Kinesio Taping and compression stockings on pain, edema, functional capacity and quality of life in patients with chronic venous disease: a randomized controlled trial. Clin Rehabil. 2020 Jun;34(6):783-793. doi: 10.1177/0269215520916851. Epub 2020 Apr 29. PMID 32349528
- [Background] Nishimura Y, Onoe H, Morichika Y, Perfiliev S, Tsukada H, Isa T. Time-dependent central compensatory mechanisms of finger dexterity after spinal cord injury. Science. 2007 Nov 16;318(5853):1150-5. doi: 10.1126/science.1147243. PMID 18006750